CLINICAL TRIAL: NCT02664155
Title: Venous Thromboembolism in Renally Impaired Patients and Direct Oral Anticoagulants
Acronym: VERDICT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: recruiting difficulties
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1508189; 2016-000858-35 (EudraCT Number)
Record Dates: First submitted 2016-01-22; First posted 2016-01-26 (Estimated); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Renal Insufficiency
Keywords: Renal insufficiency; Direct oral anticoagulants (DOA); Deep Vein Thrombosis (DVT); Pulmonary Embolism (PE); Venous Thromboembolism (VTE); Heparins
MeSH Terms: conditions — Renal Insufficiency; Venous Thrombosis; Pulmonary Embolism; Venous Thromboembolism | interventions — apixaban; Rivaroxaban; Heparin; acarboxyprothrombin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DOA : Direct Oral Anticoagulants (Experimental): The experimental group receiving DOA regimens: patients will be secondarily randomly assigned within DOAs group between:
  * Apixaban (Eliquis® tablet) 10 mg bid for 7 days then 2.5 mg bid for 3 months
  * Rivaroxaban (Xarelto® tablet) 15 mg bid for 21 days then 15 mg od for 3 months.
  Interventions: Drug: Apixaban; Drug: Rivaroxaban
- SOC : Standard Of Care (Active Comparator): The control group receiving the standard of care (SOC), i.e. heparins/VKA regimen. Patients will receive the current recommended therapy: subcutaneous or intravenous UFH/VKA in case of severe renal insufficiency and subcutaneous LMWH/VKA in case of moderate renal insufficiency for at least 5 days. VKA will begin concomitantly and continue for 3 months.
  Interventions: Drug: Heparin; Drug: VKA

INTERVENTIONS:
Drug: Apixaban — Direct Oral Anticoagulant
  Other Names: Eliquis®
  Arms: DOA : Direct Oral Anticoagulants
Drug: Rivaroxaban — Direct Oral Anticoagulant
  Other Names: Xarelto®
  Arms: DOA : Direct Oral Anticoagulants
Drug: Heparin — Standard Of Care
  Arms: SOC : Standard Of Care
Drug: VKA — Standard Of Care
  Other Names: vitamin K antagonists
  Arms: SOC : Standard Of Care

SUMMARY:
In renally impaired patients with acute venous thromboembolism (VTE), standard-of-care (SOC) anticoagulation, i.e. heparins-vitamin K antagonists (VKA), at therapeutic dosage is associated with an increased risk of thromboembolic and bleeding complications compared to patients with normal renal function. Direct oral anticoagulants (DOAs) have been shown to be at least as effective and safe as SOC in VTE treatment. But in the clinical trials, moderate renally impaired patients were poorly represented and patients with severe renal insufficiency not at all. So no dose reduction was considered.

Surprisingly, DOAs have been approved for VTE treatment in moderate and severe renally impaired patients. There is need to evaluate a reduced dose of DOAs for VTE treatment in patients with moderate and severe renal insufficiency.

We plan to evaluate reduced doses of 2 DOAs (apixaban, rivaroxaban) compared to SOC in VTE patients with moderate or severe renal insufficiency in terms of net clinical benefit (recurrent VTE and major bleeding) at 3 months.

DETAILED DESCRIPTION:
In renally impaired patients with acute venous thromboembolism (VTE), standard-of-care (SOC) anticoagulation, i.e. heparins-vitamin K antagonists (VKA), at therapeutic dosage is associated with an increased risk of thromboembolic and bleeding complications compared to patients with normal renal function. These patients represent more than 20% of the VTE population in clinical practice. Direct oral anticoagulants (DOAs) have been shown to be at least as effective and safe as SOC in VTE treatment. But in the clinical trials, moderate renally impaired patients were poorly represented (<10%) and patients with severe renal insufficiency not at all. So no dose reduction was considered.

The new DOAs have also been developed for stroke prevention in atrial fibrillation (SPAF). Patients including in AF trials are generally older and more prone to present renal impairment (>20%) than in VTE trials. So a reduced dose of DOAs was evaluated and shown to be at least as effective as, and safer than VKA in the subgroup of patients with moderate renal insufficiency (creatinine clearance between 30 to 50 ml/min).

Surprisingly, DOAs have been approved for VTE treatment and SPAF in moderate and severe renally impaired patients (creatinine clearance between 15 to 30 mL/min). Moreover, patients have to receive a reduced dose of DOAs for SPAF but a full dose of DOAs for VTE that could be associated with an increased bleeding risk, as suggested by some subgroup analyses. So, there, there is need to evaluate a reduced dose of DOAs for VTE treatment in patients with moderate and severe renal insufficiency (creatinine clearance between 15 to 50 mL/min).

Apixaban and rivaroxaban appear to be the best candidates since:

* both are approved in France in VTE patients
* they have mixed pathway of elimination (hepatic and renal)
* they have several other pharmacological similarities and they respective clinical trials have shown similar efficacy and safety profiles when compared with SOC for VTE treatment.
* they do not need to be preceded by initial parenteral heparins on the contrary to dabigatran and edoxaban. This allows evaluating the impact of DOAs in renally impaired patients independently from the initial heparins effect
* a reduced dose regimen is available and approved in AF
* the evaluation of 2 DAOs allows evaluating the concept of this new class in renally impaired VTE patients independently from the pharmaceutical companies.

Finally we plan to evaluate reduced doses of 2 DOAs (apixaban, rivaroxaban) compared to SOC in VTE patients with moderate or severe renal insufficiency in terms of net clinical benefit (recurrent VTE and major bleeding) at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a moderate renal insufficiency defined by a creatinine clearance between 30 to 50 ml/min (Cockcroft and Gault formulae) or a severe renal insufficiency (between 15 to 29 ml/min)
* Patients with acute objectively confirmed symptomatic proximal deep-vein thrombosis (DVT) or pulmonary embolism (PE) (with or without deep-vein thrombosis), planned to be treated for at least 3 months
* Patients >18 years
* Life expectancy more than 3 months
* Social security affiliation
* Signed informed consent

Exclusion Criteria:

* Indication for anticoagulants other than VTE
* Active bleeding or a high risk of bleeding contraindicating anticoagulant treatment; a systolic blood pressure of more than 180 mm Hg or a diastolic blood pressure of more than 110 mm Hg
* Anticoagulation for more than 72 hours prior to randomization
* Chronic liver disease or chronic hepatitis
* Patient at high risk of bleeding
* Creatinine clearance <15 ml/min or end stage renal disease or indication for extra-renal dialysis
* Need for concomitant anti-platelet therapy other than aspirin 75-325 mg per day. However concomitant treatment with aspirin is discouraged in this population at bleeding risk.
* Concomitant use of a strong inhibitor of cytochrome P-450 3A4 (CYP3A4) (e.g., a protease inhibitor for human immunodeficiency virus infection or azole-antimycotics agents ketoconazole, itraconazole, voriconazole, posaconazole) or a CYP3A4 inducer (e.g., rifampin, carbamazepine, or phenytoin),
* Active pregnancy or expected pregnancy or no effective contraception
* Any contraindication listed in the local labeling of UFH, LMWH or VKA or oral anticoagulant.
* Cancer-associated VTE requiring long-term treatment with LMWH
* Life expectancy of less than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2016-10-19 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Non inferiority of reduced doses of DOAs | Month 3
  To demonstrate that reduced doses of DOAs (rivaroxaban or apixaban) are non-inferior to standard of care (heparins/VKA) on the net clinical benefit (recurrent VTE and major bleeding) in renally impaired patients suffering from an acute VTE.

SECONDARY OUTCOMES:
Bleeding events | Month 3
  To demonstrate the non--inferiority of reduced dose of DOAs on the risk of major bleedings.
Venous Thromboembolism (VTE) events | Month 3
  To demonstrate the non--inferiority of reduced dose of DOAs on the risk of recurrent VTE.

CONTACTS AND LOCATIONS:
Overall Officials: MISMETTI Patrick, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (31):
- France (31):
  - CH ARRAS, Arras, Boulevard Georges Besnier
  - Chu Tours, Tours, Hôpital Trousseau
  - CH d'Agen-Nérac, Agen
  - Chu Amiens, Amiens
  - Chu Angers, Angers
  - CH Besançon, Besançon
  - CHU de Bordeaux, Bordeaux
  - CHU La Cavale Blanche Brest, Brest
  - HIA de Brest, Brest
  - CHU Castelnau-le-Lez, Castelnau-le-Lez
  - CH Louis Pasteur - Chartres, Chartres
  - Chu Clermont-Ferrand, Clermont-Ferrand
  - CHU Dijon, Dijon
  - Hôpital La Tronche Grenoble, Grenoble
  - Hôpital Charles Foix - APHP Ivry sur Seine, Ivry-sur-Seine
  - Chu Limoges, Limoges
  - CHU Lyon, Lyon
  - HCL - Hôpital Edouard Herriot, Lyon
  - Chu Montpellier, Montpellier
  - CHU de Nantes - Hôpital Bellier, Nantes
  - CHU de Nantes - Hôpital Hôtel Dieu, Nantes
  - CHU Nice, Nice
  - HEGP - APHP Paris, Paris
  - Hôpital Louis Mourier- APHP Paris, Paris
  - CHU de Rouen, Rouen
  - Chu Saint Etienne, Saint-Etienne
  - Chu Strasbourg, Strasbourg
  - CH Toulon, Toulon
  - HIA de Toulon, Toulon
  - CHU Toulouse, Toulouse
  - CH de Valenciennes, Valenciennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wetmore JB, Herzog CA, Yan H, Reyes JL, Weinhandl ED, Roetker NS. Apixaban versus Warfarin for Treatment of Venous Thromboembolism in Patients Receiving Long-Term Dialysis. Clin J Am Soc Nephrol. 2022 May;17(5):693-702. doi: 10.2215/CJN.14021021. Epub 2022 Apr 25. PMID 35470214